CLINICAL TRIAL: NCT07276581
Title: A Multicentre, Parallel-group, Phase II, Randomised, Double-blind, 4 Arm Study to Evaluate Efficacy and Safety of AZD1163 in Participants With Moderately-to-Severely Active Rheumatoid Arthritis (LaunchPAD-RA)
Brief Title: A Study to Investigate Efficacy and Safety of AZD1163 in Participants With Rheumatoid Arthritis
Acronym: LaunchPAD-RA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9640C00003; 2025-522076-85 (Other: EU CT number); 167070 (Registry Identifier: IND)
Record Dates: First submitted 2025-12-01; First posted 2025-12-11 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; AZD1163; placebo-controlled; double-blind; csDMARDs; TNFi; PAD2/4 inhibitor
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AZD1163 Dose 1 (Experimental): Participants will receive subcutaneous (SC) injection of AZD1163 Dose 1 in combination with SoC (csDMARDs or TNFi +/- csDMARD) until Week 24.
  Interventions: Drug: AZD1163
- AZD1163 Dose 2 (Experimental): Participants will receive SC injection of AZD1163 Dose 2 in combination with SoC (csDMARDs or TNFi +/- csDMARD) until Week 24.
  Interventions: Drug: AZD1163
- AZD1163 Dose 3 (Experimental): Participants will receive SC injection of AZD1163 Dose 3 in combination with SoC (csDMARDs or TNFi +/- csDMARD) until Week 24.
  Interventions: Drug: AZD1163
- Placebo (Placebo Comparator): Participants will receive SC injection of placebo matched with AZD1163 dose in combination with SoC (csDMARDs or TNFi +/- csDMARD) until Week 24.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AZD1163 — Participants will receive SC injection of one of three different doses of AZD1163 in combination with SoC (csDMARD or TNFi +/- csDMARDSoC) until Week 24.
  Arms: AZD1163 Dose 1; AZD1163 Dose 2; AZD1163 Dose 3
Other: Placebo — Participants will receive SC injection of placebo matched to AZD1163 in combination with SoC (csDMARD or TNFi +/- csDMARDSoC) until Week 24.
  Arms: Placebo

SUMMARY:
Phase II study in participants with moderately-to-severely active rheumatoid Arthritis (RA) to evaluate efficacy and safety of AZD1163.

DETAILED DESCRIPTION:
AZD1163 is a novel bispecific antibody that inhibits the activity of extracellular peptidyl arginine deiminase 2 (PAD2) and peptidyl arginine deiminase 4 (PAD4) enzymes, which are responsible for protein citrullination. In RA, citrullinated proteins lead to the production of pathogenic anti-citrullinated peptide antibodies (ACPA).

This is a Phase II, randomised, double-blind, multicentre, 4 arm placebo-controlled study designed to evaluate the efficacy and safety of AZD1163 in ACPA + adults with moderate-to-severely active RA on standard of care (SoC) (conventional synthetic disease-modifying antirheumatic drugs [csDMARDs] or tumour necrosis factor inhibitor [TNFi] +/- csDMARD).

The study will have a screening period followed by a randomisation period wherein approximately 320 participants will be randomised in a 1:1:1:1 ratio to receive study intervention.

Participants will receive subcutaneous (SC) injection of one of three different doses of AZD1163 or placebo, along with SoC until Week 24 followed by a safety follow-up (FU) period of 28 days.

ELIGIBILITY:
* Inclusion

  * Diagnosed with adult-onset RA as defined by the 2010 ACR/EULAR classification criteria for at least 12 weeks prior to screening.
  * Moderately-to-severely active RA as defined by: a. >= 6 swollen joints on 66SJC and >= 6 tender joints on 68TJC; b. CRP > upper limit of normal.
  * Have a positive ACPA at screening.
  * A history of inadequate response, or loss of response, or intolerance to: a. at least one csDMARD treatment, AND/OR b. At least one and at most 2 TNFi.
  * A history of at least 12 weeks treatment and >= 4 weeks stable on a csDMARD and/or SC TNFi prior to the day of randomisation.
* Exclusion

  * History or evidence of an alternate autoimmune or other condition that could confound the diagnosis of RA. Participants with RA and secondary Sjogren's disease are eligible.
  * Have received or planning to receive any biologic DMARDs (except for TNFi) or targeted synthetic DMARDs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2027-11-12 (Estimated); Study Completion 2028-08-18 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Disease Activity Score-C-Reactive Protein (DAS28-CRP) at Week 12 | Week 12
  Change from baseline in DAS28-CRP at Week 12.

SECONDARY OUTCOMES:
Percentage of Participants Achieving American College of Rheumatology Response Criteria 20 (ACR20) at Week 12 | Week 12
  Proportion of participants achieving a 20% improvement in ACR response criteria at Week 12.
Percentage of Participants Achieving ACR50 at Week 12 | Week 12
  Proportion of participants achieving a 50% improvement in ACR response criteria at Week 12.
Change From Baseline in Clinical Disease Activity Index (CDAI) at Week 12 | Week 12
  Change from baseline in CDAI at Week 12.
Change From Baseline in Simplified Disease Activity Index (SDAI) at Week 12 | Week 12
  Change from baseline in SDAI at Week 12.
Summary statistics to evaluate the PK of AZD1163 | Week 0 to Week 24 and Follow-Up
  AZD1163 concentrations in serum
Summary statistics to evaluate the immunogenicity of AZD1163 | Week 0 to Week 24 and Follow-Up
  ADA (incidence, prevalence, and titres)

CONTACTS AND LOCATIONS:
Locations (103):
- United States (19):
  - Research Site, Glendale, Arizona
  - Research Site, Prescott Valley, Arizona
  - Research Site, La Jolla, California
  - Research Site, San Dimas, California
  - Research Site, Boynton Beach, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, South Miami, Florida
  - Research Site, Tampa, Florida
  - Research Site, Willowbrook, Illinois
  - Research Site, Lake Charles, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, New Bedford, Massachusetts
  - Research Site, Henderson, Nevada
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Austin, Texas
  - Research Site, Baytown, Texas
  - Research Site, Houston, Texas
  - Research Site, Mesquite, Texas
  - Research Site, Tomball, Texas
- Argentina (6):
  - Research Site, Buenos Aires
  - Research Site, Caba
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, San Isidro
  - Research Site, San Miguel de Tucumán
- Brazil (5):
  - Research Site, Juiz de Fora
  - Research Site, Pelotas
  - Research Site, Porto Alegre
  - Research Site, Salvador
  - Research Site, São Paulo
- Bulgaria (3):
  - Research Site, Haskovo
  - Research Site, Pleven
  - Research Site, Sofia
- Canada (2):
  - Research Site, Windsor, Ontario
  - Research Site, Trois-Rivières, Quebec
- Chile (6):
  - Research Site, Providencia
  - Research Site, Santiago
  - Research Site, Temuco
  - Research Site, Valdivia
  - Research Site, Victoria
  - Research Site, Viña del Mar
- China (6):
  - Research Site, Beijing
  - Research Site, Jiujiang
  - Research Site, Kunming
  - Research Site, Nanchong
  - Research Site, Panjin
  - Research Site, Pingxiang
- Germany (3):
  - Research Site, Berlin
  - Research Site, Hamburg
  - Research Site, Sendenhorst
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Gyula
  - Research Site, Szeged
  - Research Site, Székesfehérvár
  - Research Site, Veszprém
- Japan (16):
  - Research Site, Bunkyō City
  - Research Site, Fukuoka
  - Research Site, Hamamatsu
  - Research Site, Hitachi-Naka
  - Research Site, Iizuka-shi
  - Research Site, Kawachinagano-shi
  - Research Site, Matsuyama
  - Research Site, Meguro-ku
  - Research Site, Miyazaki
  - Research Site, Nagoya
  - Research Site, Okayama
  - Research Site, Sagamihara-shi
  - Research Site, Sapporo
  - Research Site, Sasebo-shi
  - Research Site, Sayama-shi
  - Research Site, Yokohama
- Mexico (8):
  - Research Site, Chihuahua City
  - Research Site, Estado de México
  - Research Site, Guadalajara
  - Research Site, Gustavo A. Madero
  - Research Site, Mexico City
  - Research Site, Mérida
  - Research Site, Monterrey
  - Research Site, San Luis Potosí City
- Poland (4):
  - Research Site, Krakow
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wroclaw
- South Africa (6):
  - Research Site, Brackenfell
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Pinelands
  - Research Site, Pretoria
  - Research Site, Stellenbosch
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Málaga
  - Research Site, Sabadell
  - Research Site, Santiago de Compostela
  - Research Site, Valencia
- Ukraine (4):
  - Research Site, Ivano-Frankivsk
  - Research Site, Kyiv
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
- United Kingdom (4):
  - Research Site, Glasgow
  - Research Site, Leeds
  - Research Site, Luton
  - Research Site, Staffordshire

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/